CLINICAL TRIAL: NCT05813548
Title: The Effectiveness of an Application-Based Lifestyle Change Program on Body Composition, Health, Body Image, and Self-Esteem in Women 30 to 55 Years Old
Brief Title: The Effectiveness on an Application-Based Lifestyle Change Program on Health in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012023
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Body Image; Self Esteem; Weight Loss; Health Behavior; Health-Related Behavior; Health Knowledge, Attitudes, Practice
Keywords: Mobile Application; Phone Application; Body Composition
MeSH Terms: conditions — Weight Loss; Health Behavior; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): FASTer Way Application-Based Lifestyle Program
  Interventions: Other: FASTer Way Intervention
- Control (Active Comparator): General health and dietary guidelines
  Interventions: Other: Control Group Intervention

INTERVENTIONS:
Other: FASTer Way Intervention — 6-weeks of exercise, building healthy nutritional habits such as intermittent fasting and carb-cycling
  Arms: Treatment
Other: Control Group Intervention — 6-weeks of following general exercise and nutrition guidelines from American Heart Association (AHA) and United States Department of Agriculture (USDA), respectively.
  Arms: Control

SUMMARY:
The purpose of this study will be to examine the effectiveness of an application-based lifestyle change program on body composition, body shape, body, image, and self-esteem in females following a 6-week period. The study will be carried out in a randomized, placebo-controlled, parallel manner. Participants will be stratified into quartiles based on their body mass indices during screening and prior to baseline testing. Participants from each quartile will be randomly divided by into experimental or control conditions.

Following randomization, participants will be baseline assessed on their body composition using a whole body Dual Energy X-Ray Absorptiometry scan, on their subjective measures of body shape and image using a variety of questionnaires, blood chemistry panel, and lower-body strength using a isometric mid-thigh pull dynamometer. Following baseline testing, participants will undergo 6-weeks of following their respective condition. Participants will be instructed to follow their group-specific guidelines for the 6-week period to the best of their ability. Body shape and image questionnaires and assessments of body composition, blood chemistry, and lower-body strength will be conducted following the week 6 to conclude the study.

DETAILED DESCRIPTION:
The purpose of this study will be to examine the effectiveness of an application-based lifestyle change program on body composition, body shape, body, image, and self-esteem in females following a 6-week period. The study will be carried out in a randomized, placebo-controlled, parallel manner. Participants will be stratified into quartiles based on their body mass indices during screening and prior to baseline testing. Participants from each quartile will be randomly divided by into experimental or control conditions.

Following randomization, participants will be baseline assessed on their body composition using a whole body Dual Energy X-Ray Absorptiometry scan, on their subjective measures of body shape and image using a variety of questionnaires, blood chemistry panel, and lower-body strength using a isometric mid-thigh pull dynamometer. Following baseline testing, participants will undergo 6-weeks of following their respective condition. Participants will be instructed to follow their group-specific guidelines for the 6-week period to the best of their ability. Body shape and image questionnaires and assessments of body composition, blood chemistry, and lower-body strength will be conducted following the week 6 to conclude the study.

Participants will be assessed for the following variables on Week 0 and 6:

Primary Variables:

• Fat-, lean-, total-mass, body fat percentage, body mass index, and visceral adipose tissue via Dual Energy X-Ray Absorptiometry (DEXA)

Subjective measures related to body shape, body image, and body acceptance by administering the the following questionnaires

* Body Image and Acceptance Action Questionnaire (BI-AAQ)
* Body Shape Questionnaire (BSQ)

Secondary Variables:

* Complete Blood Count (CBC)
* Comprehensive Metabolic Panel (CMP)
* Blood Lipid Profile
* C-Reactive Protein
* Apolipoprotein B
* Lower-body strength via Isometric Mid-Thigh Pull (IMTP)
* Blood pressure
* Resting heart rate
* Pulse wave velocity

Subjective measures related to self-esteem, physical activity, and general health by administering the the following questionnaires

* Rosenberg Self-Esteem Scale (RSE)
* Modified Huet Questionnaire
* General Healthy and Activity Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between 30 and 55 years old
* Body Mass Index (BMI) between 25 and 35 kg/m^2
* Little to no recent exercise training experience (≤ 1 day per week) within the last 6 months and no recent (≤ 3-months) musculoskeletal injuries
* Willing and able to give written informed consent
* Able to read, understand, sign and date the informed consent document (English only)
* Subjects located in the Tampa Bay area who are willing to comply with the schedule visit(s) and study requirements.
* Consistent access to a smartphone with the ability to navigate an English-language application

Exclusion Criteria:

* Diagnosed cardiovascular, neurological, metabolic, musculoskeletal, renal, pulmonary, hepatic, autoimmune, or endocrine disease
* Drink heavily (>7 and >14 drinks per week for women and men, respectively)
* Exercising greater than 1 day per week for the past 6 months
* Significant food allergies or dietary restrictions
* Pregnant, breastfeeding (≤ 3-months), or seeking to become pregnant
* Smoke
* Peptic ulcer
* Any malignancy
* Thrombosis
* Undergone surgery that affects digestion and absorption
* Hypo- or hypertensive
* Undergoing hormone replacement therapy
* Using hormone boosting supplements (herbal or synthetic)
* Using drugs that are anti-diabetic, anti-platelet, anti-coagulant, or beta blockers
* Have participated in a clinical trial within the past 6 months

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in Fat Mass | Week 0 and 6
  Total fat mass will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Lean Mass | Week 0 and 6
  Total lean mass will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Total Mass | Week 0 and 6
  Total mass will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Visceral Adipose Tissue (VAT) | Week 0 and 6
  Total VAT will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Body Fat Percentage | Week 0 and 6
  Total body fat percentage will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Body Mass Index | Week 0 and 6
  Total body mass index will be assessed via dual-energy X-ray absorptiometry (DEXA)
Changes in Body Shape | Week 0 and 6
  Assessed by administering the Body Shape Questionnaire (BSQ) for subjective measurement. Values range from 1 to 6 with lower scores demonstrating a better outcome.
Changes in Body Image Acceptance | Week 0 and 6
  Assessed by administering the Body Image and Acceptance Action Questionnaire (BI-AAQ) for subjective measurement. Values range from 1 to 7 with lower scores demonstrating a better outcome.

SECONDARY OUTCOMES:
Changes in Self-Esteem | Week 0 and 6
  Assessed by administering the Rosenberg Self-Esteem Scale (RSE) for subjective measurement. Values range from 1 to 4 with higher scores demonstrating a better outcome.
Changes in General Health | Week 0 and 6
  Assessed by administering the General Health and Activity Questionnaire for subjective measurement. Values range from 0 to 20 with higher scores demonstrating a better outcome.
Changes in Modified Huet | Week 0 and 6
  Assessed by administering the Modified Huet Questionnaire for subjective measurement. Values range from 0 to 3.5 with higher scores demonstrating a better outcome.
Changes in lower-body strength | Week 0 and 6
  Assessed using the isometric mid-thigh pull
Resting Heart Rate | Week 0 and 6
  Changes in resting heart rate
Resting Systolic Blood Pressure | Week 0 and 6
  Changes in resting systolic blood pressure
Resting Diastolic Blood Pressure | Week 0 and 6
  Changes in resting diastolic blood pressure
Resting Mean Arterial Pressure | Week 0 and 6
  Changes in resting mean arterial pressure
Resting Pulse Wave Velocity | Week 0 and 6
  Changes in pulse wave velocity
Changes in C-reactive protein | Week 0 and 6
  Experimental outcome examining the total C-reactive protein via fasted whole blood samples.
Changes in Apolipoprotein B | Week 0 and 6
  Experimental outcome examining the total Apolipoprotein B via fasted whole blood samples.
Changes in White Blood Cell count | Week 0 and 6
  Experimental outcome examining the total white blood cell count via fasted whole blood samples.
Changes in Red Blood Cell count | Week 0 and 6
  Experimental outcome examining the total red blood cell count via fasted whole blood samples.
Changes in Hemoglobin levels | Week 0 and 6
  Experimental outcome examining the total hemoglobin via fasted whole blood samples.
Changes in Hematocrit levels | Week 0 and 6
  Experimental outcome examining the total hematocrit via fasted whole blood samples.
Changes in Mean Corpuscular Volume | Week 0 and 6
  Experimental outcome examining the total mean corpuscular volume via fasted whole blood samples.
Changes in Mean Corpuscular Hemoglobin | Week 0 and 6
  Experimental outcome examining the total mean corpuscular hemoglobin via fasted whole blood samples.
Changes in Mean Corpuscular Hemoglobin Concentration | Week 0 and 6
  Experimental outcome examining the total mean corpuscular hemoglobin concentration via fasted whole blood samples.
Changes in Red Cell Distribution Width | Week 0 and 6
  Experimental outcome examining the total red cell distribution width via fasted whole blood samples.
Changes in Platelet Count | Week 0 and 6
  Experimental outcome examining the total platelet count via fasted whole blood samples.
Changes in Mean Platelet Volume | Week 0 and 6
  Experimental outcome examining the total mean platelet volume via fasted whole blood samples.
Changes in Granulocyte levels | Week 0 and 6
  Experimental outcome examining the percentage of Granulocytes via fasted whole blood samples.
Changes in Lymphocyte levels | Week 0 and 6
  Experimental outcome examining the percentage of Lymphocytes via fasted whole blood samples.
Changes in Monocyte levels | Week 0 and 6
  Experimental outcome examining the percentage of Monocytes via fasted whole blood samples.
Changes in Eosinophil levels | Week 0 and 6
  Experimental outcome examining the percentage of Eosinophil via fasted whole blood samples.
Changes in Basophil levels | Week 0 and 6
  Experimental outcome examining the percentage of Basophil via fasted whole blood samples.
Changes in Granulocyte count | Week 0 and 6
  Experimental outcome examining total Granulocytes via fasted whole blood samples.
Changes in Lymphocyte count | Week 0 and 6
  Experimental outcome examining total Lymphocytes via fasted whole blood samples.
Changes in Monocyte count | Week 0 and 6
  Experimental outcome examining total Monocytes via fasted whole blood samples.
Changes in Eosinophil count | Week 0 and 6
  Experimental outcome examining total Eosinophils via fasted whole blood samples.
Changes in Basophil count | Week 0 and 6
  Experimental outcome examining total Basophils via fasted whole blood samples.
Changes in Glucose levels | Week 0 and 6
  Experimental outcome examining total glucose via fasted whole blood samples.
Changes in Blood Urea Nitrogen levels | Week 0 and 6
  Experimental outcome examining total blood urea nitrogen via fasted whole blood samples.
Changes in Serum Creatinine levels | Week 0 and 6
  Experimental outcome examining total serum creatinine via fasted whole blood samples.
Changes in Sodium levels | Week 0 and 6
  Experimental outcome examining total sodium via fasted whole blood samples.
Changes in Potassium levels | Week 0 and 6
  Experimental outcome examining total potassium via fasted whole blood samples.
Changes in Chloride levels | Week 0 and 6
  Experimental outcome examining total chloride via fasted whole blood samples.
Changes in Carbon Dioxide levels | Week 0 and 6
  Experimental outcome examining total carbon dioxide via fasted whole blood samples.
Changes in Calcium levels | Week 0 and 6
  Experimental outcome examining total calcium via fasted whole blood samples.
Changes in Total Protein levels | Week 0 and 6
  Experimental outcome examining total Protein via fasted whole blood samples.
Changes in Albumin levels | Week 0 and 6
  Experimental outcome examining total albumin via fasted whole blood samples.
Changes in Globulin levels | Week 0 and 6
  Experimental outcome examining total globulin via fasted whole blood samples.
Changes in Total Bilirubin levels | Week 0 and 6
  Experimental outcome examining total bilirubin via fasted whole blood samples.
Changes in Alkaline Phosphate levels | Week 0 and 6
  Experimental outcome examining total alkaline phosphate via fasted whole blood samples.
Changes in Alanine Transaminase levels | Week 0 and 6
  Experimental outcome examining total Alanine Transaminase via fasted whole blood samples.
Changes in Aspartate Aminotransferase levels | Week 0 and 6
  Experimental outcome examining total Aspartate Aminotransferase via fasted whole blood samples.
Changes in Albumin to Globulin ratio | Week 0 and 6
  Experimental outcome examining the ratio of Albumin to Globulin via fasted whole blood samples.
Changes in Blood Urea Nitrogen to Creatinine ratio | Week 0 and 6
  Experimental outcome examining the ratio of Blood urea nitrogen to Creatinine via fasted whole blood samples.
Changes in estimated Glomerular Filtration Rate | Week 0 and 6
  Experimental outcome examining the Glomerular filtration rate via fasted whole blood samples.
Changes in Total Cholesterol levels | Week 0 and 6
  Experimental outcome examining total cholesterol via fasted whole blood samples.
Changes in Triglyceride levels | Week 0 and 6
  Experimental outcome examining total triglycerides via fasted whole blood samples.
Changes in High Density Lipoprotein levels (HDL) | Week 0 and 6
  Experimental outcome examining total high density lipoprotein via fasted whole blood samples.
Changes in Low Density Lipoprotein levels (LDL) | Week 0 and 6
  Experimental outcome examining total low density lipoprotein via fasted whole blood samples.
Changes in Cholesterol to High Density Lipoprotein ratio | Week 0 and 6
  Experimental outcome examining the ratio of Cholesterol to High density lipoprotein via fasted whole blood samples.
Adverse Effects | Week 0 and 6
  Defined as participants self-reported adverse effects. Items that will be surveyed are headache, dizziness, nausea, vomiting, indigestion, blurred vision, lethargy, swelling, itching, chest pain, heart palpitations, difficulty breathing, lethargy, and muscle cramps.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science and Performance Institute, Tampa, Florida, United States

REFERENCES:
- [Derived] Ottinger CR, Gheith RH, Sharp MH, Davis JM, Lowery RP, Wilson JM. A randomized controlled trial to assess the effectiveness of a mobile application-based lifestyle change program (FASTer Way) on body composition, biochemical and hematological health markers, body image, and self-esteem in overweight women. Mhealth. 2025 Mar 20;11:13. doi: 10.21037/mhealth-24-62. eCollection 2025. PMID 40248760